CLINICAL TRIAL: NCT02893813
Title: Comparison Between Two Surgical Methods for Eyelid Ectropion: Tarsal Strip Alone Versus Tarsal Strip With Punctoplasty (Three Snips With or Without Diamond-shaped Resection)
Acronym: ECTROPALP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-10Obs-CHRMT
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Ectropion
MeSH Terms: conditions — Ectropion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Ectropion of the eyelid can lead to skin retraction, stenosis of lacrimal point, chronic watering, visual discomfort or low visual acuity, mostly when it occurs with ectropion of lacrimal point. The objective of the study is to compare two surgical strategies for eyelid ectropion combined with ectropion of the lacrimal point

DETAILED DESCRIPTION:
Were included patients underwent eyelid ectropion surgery in ophthalmology department from Oct 2014 to Oct 2015. The first procedure is lateral tarsal strip alone (group 1); the second one is lateral tarsal strip with three snips with or without diamond-shaped resection (group 2). The authors focused on the alteration of the quality of life related to watering, before and after operation. Quality of life related to discomfort due to watering was evaluated before and after surgery using a questionnaire. Informations have been gathered via phone with a ten items questionnaire, each item is worth 0 (no or minim discomfort due to watering) or 1 (discomfort due to more than moderated watering)

ELIGIBILITY:
Inclusion Criteria:

* patients underwent eyelid ectropion surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent eyelid ectropion surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of life related to discomfort due to watering after eyelid ectropion surgery | 1 year
  questionnaire quality of life